CLINICAL TRIAL: NCT04531709
Title: Financial Toxicity and Quality of Life in Patients With Testicular Germ Cell Tumors
Brief Title: Financial Toxicity and Quality of Life in Patients With TGCT
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: CTMS 20-0061; HSC20200462E (Other: UT Health Science Center San Antonio IRB)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Testicular Neoplasm
MeSH Terms: conditions — Testicular Neoplasms | interventions — Costs and Cost Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-term survivors of TGCT
  Interventions: Other: Comprehensive Score for financial toxicity (COST); Other: Functional Assessment of Cancer Therapy: General (FACT-G); Other: EORTC QLQ C-30; Other: EORTC QLQ-TC26.

INTERVENTIONS:
Other: Comprehensive Score for financial toxicity (COST) — Measure indirect and direct health care cost that burden patients and their loved ones.
Other: Functional Assessment of Cancer Therapy: General (FACT-G) — General quality of life instrument
Other: EORTC QLQ C-30 — Assess quality of life in cancer patients
Other: EORTC QLQ-TC26. — To measure disease and treatment related quality of life issues relevant to testicular cancer patients that were not explored in the QLQ-C30 questionnaire.

SUMMARY:
This is a cross-sectional, observational study employing validated questionnaires to investigate financial toxicity in subjects with testicular germ cell tumors (TGCT). As background, TGCTs are the most common malignancies among men from age 15-35. Treatment is highly curative, but often consists of intensive multi-cycle chemotherapy with significant potential for physical toxicity. The treatment course itself is disruptive and long term physical and mental health consequences can increase risk for financial toxicity. Thus, we aim to study financial toxicity in both patients with TGCT actively receiving treatment and in TGCT survivors. There will be two separate cohorts: Cohort 1 will consist of subjects with recently diagnosed TGCT who will undergo multi-agent, multi-cycle chemotherapy and Cohort 2 will consist of subjects who have completed chemotherapy and are long-term survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Patients with histologically or clinically confirmed germ cell tumor.
* Completed treatment for germ cell tumor with multicycle (> 2 cycles) / multiagent chemotherapy.
* Within years 1-5 of surveillance since Day 1 of last cycle of chemotherapy
* Signed informed consent

Exclusion Criteria:

* Long-term survivors

  * Patients undergoing active chemotherapy
  * Patients who did not complete 1st line chemotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients diagnosed with testicular germ cell tumors TGCT, divided into non-seminomatous germ cell tumors (NSGCT) and seminomas; both of which are treated with a combination of surgery and chemotherapy or radiation depending on stage of disease.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Number of patients undergoing treatment for newly diagnosed GCT and GCT patients who are currently in surveillance whose levels of financial toxicity are high. | 5 years

SECONDARY OUTCOMES:
Number and type of financial risk factors impacting low levels of health-related quality of life for patients with GCT. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Pruthi, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Mays Cancer Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Souza JA, Yap BJ, Wroblewski K, Blinder V, Araujo FS, Hlubocky FJ, Nicholas LH, O'Connor JM, Brockstein B, Ratain MJ, Daugherty CK, Cella D. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. 2017 Feb 1;123(3):476-484. doi: 10.1002/cncr.30369. Epub 2016 Oct 7. PMID 27716900
- [Result] Nigam M, Aschebrook-Kilfoy B, Shikanov S, Eggener S. Increasing incidence of testicular cancer in the United States and Europe between 1992 and 2009. World J Urol. 2015 May;33(5):623-31. doi: 10.1007/s00345-014-1361-y. Epub 2014 Jul 17. PMID 25030752
- [Result] Baird DC, Meyers GJ, Hu JS. Testicular Cancer: Diagnosis and Treatment. Am Fam Physician. 2018 Feb 15;97(4):261-268. PMID 29671528
- [Result] Palumbo C, Mistretta FA, Mazzone E, Knipper S, Tian Z, Perrotte P, Antonelli A, Montorsi F, Shariat SF, Saad F, Simeone C, Briganti A, Lattouf JB, Karakiewicz PI. Contemporary Incidence and Mortality Rates in Patients With Testicular Germ Cell Tumors. Clin Genitourin Cancer. 2019 Oct;17(5):e1026-e1035. doi: 10.1016/j.clgc.2019.06.003. Epub 2019 Jun 13. PMID 31378580
- [Result] Mariotto AB, Yabroff KR, Shao Y, Feuer EJ, Brown ML. Projections of the cost of cancer care in the United States: 2010-2020. J Natl Cancer Inst. 2011 Jan 19;103(2):117-28. doi: 10.1093/jnci/djq495. Epub 2011 Jan 12. PMID 21228314
- [Result] Sztankay M, Aaronson NK, Arraras JI, Basso U, Bumbasirevic U, Efficace F, Giesinger JM, Johnson CD, van Leeuwen M, Oberguggenberger AS, Sosnowski R, Young T, Holzner B; European Organisation for Research and Treatment of Cancer Quality of Life Group (EORTC QLG). International phase IV validation study of an EORTC quality of life questionnaire for testicular cancer patients: the EORTC QLQ-TC26. BMC Cancer. 2018 Nov 12;18(1):1104. doi: 10.1186/s12885-018-5036-8. PMID 30419889